CLINICAL TRIAL: NCT07346339
Title: The Effect of Sensory Mindfulness Technique on Breast Milk, Maternal Well-Being, and Stress Levels in Mothers Whose Infants Are Undergoing Treatment in the Neonatal Intensive Care Unit and Are Breastfeeding With Expressed Breast Milk
Brief Title: Sensory Mindfulness for NICU Mothers: Effects on Breast Milk, Well-Being, and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Emel Yürük, Doctoral instructor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Çukurova U Ethics Commit 19/42
Record Dates: First submitted 2025-06-13; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Newborn Diseases; Breast Milk Collection; Well-being; MİNDFULNESS
Keywords: Breast milk; well-being; MİNDFULNESS
MeSH Terms: conditions — Breast Milk Expression | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: 1. Mindfulness Group
     * Mothers are informed about the study and verbal consent is obtained.
     * Written consent is obtained using the informed consent form (Appendix 1).
     * The introductory information form is completed.
     * The Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
     * Training on effective breastfeeding techniques is provided to the mother.
     * Mindfulness training is provided to the mother.
     * The mother is given a hat that her baby has worn for a while.
     * The mother is asked to smell the hat while breastfeeding, visualize her baby, look at a picture of her baby, and practice positive thinking techniques.
     * The mother records the amount of breast milk expressed and the duration of expression after each session in the observation form.
     * The mother performs this practice for the next three breastfeeding sessions and records the results.
     * After three breastfeeding sessions, the Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
  2. Control Group - Mother
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): 1. Mindfulness Group
  * Mothers are informed about the study and verbal consent is obtained.
  * Written consent is obtained using the informed consent form (Appendix 1).
  * The introductory information form is completed.
  * The Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
  * Training on effective breastfeeding techniques is provided to the mother.
  * Mindfulness training is provided to the mother.
  * The mother is given a hat that her baby has worn for a while.
  * The mother is asked to smell the hat while breastfeeding, visualize her baby, look at a picture of her baby, and practice positive thinking techniques.
  * The mother records the amount of breast milk expressed and the duration of expression after each session in the observation form.
  * The mother performs this practice for the next three breastfeeding sessions and records the results.
  * After three breastfeeding sessions, the Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
  Interventions: Behavioral: Mindfulness
- Control Group (No Intervention): * Mothers are informed about the study and verbal consent is obtained.
  * Written consent is obtained using an informed consent form.
  * The Demographic Information Form is completed.
  * The Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
  * The mother is provided with training on effective breastfeeding techniques.
  * The mother records the amount of breast milk expressed and the duration of each pumping session in the application observation form after each pumping session.
  * The mother performs this procedure for the next 3 pumping sessions and records the results.
  * The Well-Being Scale and the YYBÜ Parent Stress Scale are completed after the 3 pumping sessions.

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness Group
  * Mothers are informed about the study and verbal consent is obtained.
  * Written consent is obtained using the informed consent form (Appendix 1).
  * The introductory information form is completed.
  * The Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
  * Training on effective breastfeeding techniques is provided to the mother.
  * Mindfulness training is provided to the mother.
  * The mother is given a hat that her baby has worn for a while.
  * The mother is asked to smell the hat while breastfeeding, visualize her baby, look at a picture of her baby, and practice positive thinking techniques.
  * The mother records the amount of breast milk expressed and the duration of expression after each session in the observation form.
  * The mother performs this practice for the next three breastfeeding sessions and records the results.
  * After three breastfeeding sessions, the Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
  Arms: Mindfulness

SUMMARY:
Breast milk, which contains all the nutrients a baby needs, not only nourishes the baby but also provides many benefits for both the mother and the baby. During the first 6 months of life, breast milk is the only food that provides the energy a baby needs, supports growth and development, is easily digestible, and can be delivered to the baby without contamination due to its ready-to-use nature. Babies who are breastfed are less likely to experience oral and dental problems in later life. Breast milk strengthens the baby's immune system, protecting against conditions such as sepsis, gastroenteritis, food allergies, rhinitis, obesity, and necrotizing enterocolitis.

Mothers who breastfeed their babies are less likely to experience postpartum uterine bleeding, infection, stress, and depression. Breastfeeding mothers have a lower risk of developing diseases such as breast and ovarian cancer, osteoporosis, and cardiovascular diseases compared to non-breastfeeding mothers. On the other hand, the comfort of breastfeeding and its economic accessibility are among its other benefits. Considering all these benefits of breast milk, the United Nations Children's Fund (UNICEF) and the World Health Organization (WHO) recommend that infants be be exclusively breastfed for the first six months of life, continue breastfeeding with complementary foods after six months, and continue breastfeeding until the age of two years.

However, most premature infants are not mature enough to suckle or are admitted to the neonatal intensive care unit and therefore cannot be directly breastfed. For this reason, mothers should express their breast milk and provide it to the newborn until the infant is ready to breastfeed. However, research findings show that many mothers stop expressing milk within the first few weeks due to a decrease in milk supply, which hinders successful breastfeeding.

Various hypotheses exist regarding the decrease in milk production, including not starting to express milk early enough after birth (it is recommended to start within the first 6-12 hours); not expressing milk frequently enough (it is recommended to express every 2-3 hours to support the development of adequate milk production); not consuming enough fluids and not getting enough rest, and not feeling psychologically adequate. Some mothers need to express milk for weeks or months without skin-to-skin contact with their babies. Therefore, in addition to educational support, emotional support is also important for mothers whose babies are in the neonatal intensive care unit.

Therefore, the difficulties experienced by mothers may also affect milk production in breastfeeding mothers. Today, mindfulness-based programs are used to increase women's awareness and stress tolerance during pregnancy and the postpartum period.

Mindfulness refers to conscious awareness and can be defined as a state of consciousness that aims to focus attention on the present moment. It also involves staying connected with one's own emotions, observing what is happening around with awareness, and accepting life's experiences objectively without judgment.

Over the past decade, interest in mindfulness has grown as an increasing number of health professionals have shown interest in learning mindfulness techniques and integrating them into their therapeutic work. Studies have shown that mindfulness techniques reduce stress levels in mothers and increase breast milk volume, pumping duration, and frequency. However, the effectiveness of these techniques has been found to be dose-dependent. According to the results of a study investigating the effects of mindfulness practices in breastfeeding mothers, mothers who practiced meditation for two hours a day for eight weeks with guidance showed a decrease in anxiety and stress levels, while self-compassion and awareness levels increased significantly. In a study conducted by Massa and colleagues, the breast milk production of mothers who practiced mindfulness-based meditation and provided breast milk to preterm infants was compared with that of mothers who breastfed routinely. The results of the study revealed that mothers who meditated more frequently experienced easier milk expression and reduced symptoms of depression.

Studies show that mindfulness benefits breastfeeding and milk-expressing mothers. Breast milk also supports newborn recovery and shortens NICU stay. However, no research has yet explored sensory mindfulness in NICU mothers feeding with expressed milk.

ELIGIBILITY:
1. Mindfulness Group

   * Mothers are informed about the study and verbal consent is obtained.
   * Written consent is obtained using the informed consent form (Appendix 1).
   * The introductory information form is completed.
   * The Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
   * Training on effective breastfeeding techniques is provided to the mother.
   * Mindfulness training is provided to the mother.
   * The mother is given a hat that her baby has worn for a while.
   * The mother is asked to smell the hat while breastfeeding, visualize her baby, look at a picture of her baby, and practice positive thinking techniques.
   * The mother records the amount of breast milk expressed and the duration of expression after each session in the observation form.
   * The mother performs this practice for the next three breastfeeding sessions and records the results.
   * After three breastfeeding sessions, the Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
2. Control Group

   * Mothers are informed about the study and verbal consent is obtained.
   * Written consent is obtained using an informed consent form.
   * The Demographic Information Form is completed.
   * The Well-Being Scale and the YYBÜ Parent Stress Scale are completed.
   * The mother is provided with training on effective breastfeeding techniques.
   * The mother records the amount of breast milk expressed and the duration of each pumping session in the application observation form after each pumping session.
   * The mother performs this procedure for the next 3 pumping sessions and records the results.
   * The Well-Being Scale and the YYBÜ Parent Stress Scale are completed after the 3 pumping sessions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-09-30 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
WHO (Five) Well-Being Index | 1 months
  A short and practical measure developed by the World Health Organization to assess individuals' general well-being and quality of life.
Parental Stressor Scale | 1 months
  Parent Stress Scale (Parental Stressor Scale: Neonatal Intensive Care Unit, PSS:NICU)

CONTACTS AND LOCATIONS:
Locations (1):
- Balcalı Hastanesi, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No